CLINICAL TRIAL: NCT00525967
Title: Switching From Morphine to Oral Methadone Plus Acetaminophen in the Treatment of Cancer Pain: A Randomized, Double-Blind Study
Brief Title: Switching From Morphine to Oral Methadone Plus Acetaminophen in the Treatment of Cancer Pain
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 217/2005
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2007-09-06 (Estimated); Status verified 2007-09

CONDITIONS: Cancer; Pain; Palliative Care
Keywords: Cancer Pain; Methadone; Morphine; Acetaminophen; Palliative Care
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain | interventions — Methadone; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Methadone plus Placebo
  Interventions: Drug: Methadone plus Acetaminophen or Placebo
- 2 (Experimental): Methadone plus Acetaminophen
  Interventions: Drug: Methadone plus Acetaminophen or Placebo

INTERVENTIONS:
Drug: Methadone plus Acetaminophen or Placebo — Methadone bid according to a established conversion morphine-to-methadone ratio plus Placebo or Acetaminophen qid

SUMMARY:
The purpose of this study is to determine whether oral methadone plus acetaminophen can substitute morphine in the treatment of cancer pain.

DETAILED DESCRIPTION:
Opioids are the mainstay of moderate-to-severe cancer pain management. Although morphine is the most commonly used, methadone has some advantages such as higher potency, lower cost and longer administration intervals. To minimize the time necessary to achieve the equianalgesic effect after a switching from morphine to methadone, acetaminophen was added in the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cancer pain
* Regular use of oral Morphine

Exclusion Criteria:

* Use of Acetaminophen in the last 48 hours
* Renal or Hepatic failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-02; Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity and time to equianalgesic effect | within the first 7 days after switching

SECONDARY OUTCOMES:
Degree of nausea, vomiting, obstipation, xerostomia and drowsiness | within the first 7 days of switching

CONTACTS AND LOCATIONS:
Overall Officials: Daniel IG Cubero, Principal Investigator — Faculdade de Medicina do ABC; Auro del Giglio, Study Director — Faculdade de Medicina do ABC
Locations (1):
- Disciplina de Oncologia, Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil

REFERENCES:
- [Result] Ripamonti C, Groff L, Brunelli C, Polastri D, Stavrakis A, De Conno F. Switching from morphine to oral methadone in treating cancer pain: what is the equianalgesic dose ratio? J Clin Oncol. 1998 Oct;16(10):3216-21. doi: 10.1200/JCO.1998.16.10.3216. PMID 9779694
- [Result] Mercadante S, Casuccio A, Fulfaro F, Groff L, Boffi R, Villari P, Gebbia V, Ripamonti C. Switching from morphine to methadone to improve analgesia and tolerability in cancer patients: a prospective study. J Clin Oncol. 2001 Jun 1;19(11):2898-904. doi: 10.1200/JCO.2001.19.11.2898. PMID 11387363
- [Result] Mercadante S, Casuccio A, Calderone L. Rapid switching from morphine to methadone in cancer patients with poor response to morphine. J Clin Oncol. 1999 Oct;17(10):3307-12. doi: 10.1200/JCO.1999.17.10.3307. PMID 10506634
- [Result] Mercadante S, Ferrera P, Villari P, Casuccio A. Rapid switching between transdermal fentanyl and methadone in cancer patients. J Clin Oncol. 2005 Aug 1;23(22):5229-34. doi: 10.1200/JCO.2005.13.128. PMID 16051965
- [Result] Bruera E, Palmer JL, Bosnjak S, Rico MA, Moyano J, Sweeney C, Strasser F, Willey J, Bertolino M, Mathias C, Spruyt O, Fisch MJ. Methadone versus morphine as a first-line strong opioid for cancer pain: a randomized, double-blind study. J Clin Oncol. 2004 Jan 1;22(1):185-92. doi: 10.1200/JCO.2004.03.172. PMID 14701781
- [Result] Stockler M, Vardy J, Pillai A, Warr D. Acetaminophen (paracetamol) improves pain and well-being in people with advanced cancer already receiving a strong opioid regimen: a randomized, double-blind, placebo-controlled cross-over trial. J Clin Oncol. 2004 Aug 15;22(16):3389-94. doi: 10.1200/JCO.2004.09.122. PMID 15310785
- [Result] Mercadante S, Casuccio A, Agnello A, Serretta R, Calderone L, Barresi L. Morphine versus methadone in the pain treatment of advanced-cancer patients followed up at home. J Clin Oncol. 1998 Nov;16(11):3656-61. doi: 10.1200/JCO.1998.16.11.3656. PMID 9817288
- See also: Newsletter, March 2004 — http://www.palliativedrugs.com